CLINICAL TRIAL: NCT05084430
Title: A Phase I/II Study of Pembrolizumab and M032 (NSC 733972), a Genetically Engineered HSV-1 Expressing IL-12, in Patients With Recurrent/Progressive and Newly Diagnosed Glioblastoma Multiforme, Grade 3 or Grade 4 Astrocytoma, or Gliosarcoma
Brief Title: Study of Pembrolizumab and M032 (NSC 733972)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, James Markert, MD, Chair, Department of Neurosurgery, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300007756; 58006 (Other Grant/Funding Number: MERCK SHARP & DOHME CORP)
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma Multiforme; Anaplastic Astrocytoma; Gliosarcoma
Keywords: Recurrent; Progressive; M032; Pembrolizumab
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Gliosarcoma; Recurrence | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Recurrent Newly Diagnosed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Recurrent MG (Experimental): To determine the safety and tolerability of M032 at the doses examined when given in combinations with pembrolizumab in patients with recurrent MG.
  Interventions: Drug: M032; Drug: Pembrolizumab
- Newly Diagnosed MG (Experimental): To determine Overall Survival at 12 and 24 months, and Progression Free Survival at 6 months (PFS-6) in patients with newly diagnosed glioblastoma multiforme of M032 when given in combinations with pembrolizumab (while maintaining safety).
  Interventions: Drug: M032; Drug: Pembrolizumab

INTERVENTIONS:
Drug: M032 — Starting at week four, patients will undergo treatment on the same day, and every three weeks thereafter, with intravenous infusion of 200mg of Pembrolizumab . A total of 3 combined doses of Pembrolizumab and M032 will be given.
Drug: Pembrolizumab — Starting at week four, patients will undergo treatment on the same day, and every three weeks thereafter, with intravenous infusion of 200mg of Pembrolizumab . A total of 3 combined doses of Pembrolizumab and M032 will be given.

SUMMARY:
This Phase I (Cohort I and Cohort II) and Phase II trial is designed to confirm the safety and tolerability of Pembrolizumab when given in conjunction with M032, an Oncolytic Herpes Simplex Virus (oHSV) that expresses IL-12 and perform the Phase II portion using a Recommended Phase 2 Dose (RP2D) of M032 (provided by the Phase I) when given in conjunction with Pembrolizumab for recurrent malignant glioma (glioblastoma multiforme, anaplastic astrocytoma, or glio-sarcoma).

DETAILED DESCRIPTION:
Phase I/Cohort I:

For the Phase I portion of this trial, patients whose malignant gliomas recur after undergoing initial surgical resection, standard of care radiotherapy (60Gy) and standard of care temozolomide chemotherapy and who are candidates for, and would bene-fit from, a surgical debulking. Patients whose tumors have unmethylated MGMT promoters who have completed radiation therapy will also be eligible, regardless of whether or not they received temozolomide, since some centers are not using temozolomide in these patients. M032 will initially be administered directly into the tumor bed at the time of craniotomy and immediately after resection of the tumor. Patients will be treated with a total dose of 1 x 106 pfu of M032 initially and then subsequently with each dose of Pembrolizumab. If one toxicity occurs at a given dose level, that cohort will be increased to six patients. If two or more toxicities occur at the 1 x 106 pfu dose level, then a new cohort will be enrolled at 1 x 105 pfu, using the same approach. If two or more toxicities occur at the 1 x 105 pfu dose level, then the Data Safety and Monitoring Board (DSMB) will be consulted to determine if a stopping rule should be invoked or consideration of dose de-escalation to 1 x 104 pfu be considered. The highest safe dose will be considered the starting dose for

Phase I/Cohort II. Details of initial dose administration of M032. Patients must be candidates for a resection of the enhancing portion of the recurrent tumor; they will undergo craniotomy, with additional burr holes as needed, and then stereotactic placement of up to 4 infusion catheters. Planned catheter tip locations will include: a) > 2.5 cm from a cortical surface; b) > 1 cm from an ependymal surface or the margin of the planned resection cavity; and c) if possible, > 0.5 cm from a sulcus. This will minimize loss of dose into the subarachnoid or intra-ventricular space during subsequent M032 inoculations.

Only after catheters have been successfully placed (with Rickham reservoirs used to cap off catheters and hold them in place for the remainder of surgery) will patients will then undergo resection of the enhancing portion of the tumor. Subsequent to the resection but prior to dural closure, M032 will be administered if no ventricular entry has occurred during the resection. M032 will be administered by by multiple free hand injections into the resected tumor bed, using approximately equal volumes at each site (6 ml total). Each inoculation will be administered ~1 cm apart and delivered into the resected tumor bed over 1 minute and at a 1 cm depth (28G, 1/2-inch needle fitted to a 1-cc tuberculin syringe), where possible. Injections will be placed with careful avoidance of penetration of the ventricular system or any significant vascular structures, and any of the already-placed catheters. Intraoperative ultrasound will be used as needed to define positions of structures or catheters to avoid. After each inoculation the needle will be left in place for up to two minutes before removal and, after removal, the entry site will be covered with hemostatic agent. Both of these measures should minimize reflux of inoculum back into the tumor cavity. Before closing the dura, a fifth catheter will be left in place and then anchored with a Rickham in the tumor resection cavity to allow later access for CSF collection. This Rickham will not be used for M032 administration. The surgical procedure will then be completed in standard fashion. If ventricular entry has occurred during surgery, no M032 will be administered intraoperatively. Instead, a post-operative CT scan will be obtained on Day 1, and the initial M032 dose will be administered as outlined below, using all catheters felt to be appropriately positioned adjacent to the tumor cavity without violating the constraints of the exclusion criteria.

Pembrolizumab treatment and subsequent treatments of M032. Starting at week four, patients will undergo treatment on the same day, and every three weeks thereafter, with intra-venous infusion of 200mg of Pembrolizumab (for dosing detail, see Section 5.2.1). A total of 3 combined doses of Pembrolizumab and M032 will be given. Patients will then undergo treatment with inoculation of the calculated total dose of M032 as follows: each total dose (1 x 105 pfu for dose level one, 1 x 106 pfu for dose level two) directly into the remaining tumor bed at the time of craniotomy and immediately after resection for a particular dose level will be divided into up to four aliquots depending on the number of catheters available for inoculation. Each aliquot will be 1ml in total volume, consisting of 0.5 ml of M032 and will be infused over two minutes after puncture of each individual reservoir with a 22-24 g needle (using sterile techniques, after sterile preparation of the overlying scalp), followed by 0.5 ml of preservative free saline.

Determination of the suitability of each reservoir/catheter for inoculation will be made by the PI before each dosing and will include known patency status of each catheter, location of catheter tip and degree of adherence to the placement guidelines described above; 3) concerns for associated neurotoxicity related to M032 and/or inflammation in area of a particular reservoir/catheter tip; and 4) availability of other catheters for inoculation. Catheters whose reservoir(s) are closely associated with overlying scalp infections/inflammation will not be injected. Each catheter will be gently aspirated after the Rickham has been accessed but prior to M032 inoculation; catheters from which CSF can be aspirated will not be inoculated to avoid inoculation into the CSF space. The MRI obtained immediately prior to assessment (see schedule, below) will be used to help inform the decision-making above. If there is any question regarding reservoir/catheter suitability, an additional CT or MRI may be obtained prior to inoculation at the PI's discretion.

Combined Pembrolizumab and M032 treatments at each dose level will be repeated at three-week intervals for up to three cycles total, or until unacceptable toxicity or tumor progression occurs. Patients who are responding to treatment may be considered for additional dosing after the trial period has been completed.

The first two patients treated will not require any waiting period between enrollments. If one of the two should develop a toxicity, the third and subsequent (up to six) patients at that level will not be enrolled until seven weeks from the initial dose of M032 and three weeks from the first combined dose of Pembrolizumab and M032 has transpired for the initial two patients and every patient thereafter, to allow adequate duration of time for development of potential dose limiting toxicities in each treated patient before treating the next patient at that level.

Patients will undergo and then subsequently with each dose of Pembrolizumab; i If one toxicity occurs at a given dose level, that cohort will be increased to 6 patients. If 2 or more toxicities occur at the tested dose level, then with the approval of the DSMB, the dose will be de-escalated by one log and a new cohort enrolled with similar rules at the level. If 2 or more toxicities occur at the de-escalated dose level, then the DSMB will be consulted to determine if a stopping rule should be invoked or consideration of further dose de-escalation should be considered. The investigators anticipate as few as four patients (given two or more DLTs initially) and as many as 12 (only one DLT at each dose level). However, based on experience with M032 and Pembrolizumab, the investigators expect that this combination will not pro-duce any dose-limiting toxicities (DLTs).

Phase I/Cohort II: Having established for the safety and tolerability of M032 in conjunction with Pembrolizumab in patients with recurrent Malignant Glioma (MG), the trial will immediately transition into a Phase I Cohort II study of Pembrolizumab and M032 in patients with newly diagnosed MG. Patients who are previously untreated but suspected of having a high grade glioma by MRI and are eligible for craniotomy and resection will be offered participation in this two-Cohort trial. As in Phase I Cohort I, for the Phase I/Cohort II, consented subjects will have safe gross total resection, implantation of up to four Rickham catheters in the peritumoral brain and M032 injected into the wall of the resection cavity as described above.

Patients will be treated with a total dose of of M032 initially at the time of craniotomy as determined in Cohort I, above. They will then undergo treatment with standard fractionated radiation, and temozolomide as determined by treating physician. Starting at week four, patients will undergo treatment on the same day, and every three weeks thereafter, with intra-venous infusion of 200mg of Pembrolizumab (for dosing detail, see Section 5.2.1) and intratumoral M032 (via the Rickham-catheters placed at the periphery of the tumor cavity-the catheter left in the tumor cavity itself will not be used for M032 inoculation, but only to access CSF). Patients will then undergo treatment with inoculation of the calculated total dose of M032 for that dose level divided into up to four aliquots depending on the number of catheters available for inoculation. Each aliquot will be 1ml in total volume, consisting of 0.5 ml of M032 and will be infused over 2 minutes after puncture of each individual reservoir with a 22-24 g needle (using sterile techniques, after sterile preparation of the over-lying scalp).

Determination of the suitability of each reservoir/catheter for inoculation will be made by the PI before each dosing and will include known patency status of each catheter, location of catheter tip and degree of adherence to the placement guidelines described above; 3) concerns for associated neurotoxicity related to M032 and/or inflammation in area of a particular reservoir/catheter tip; and 4) availability of other catheters for inoculation. Catheters whose reservoir(s) are closely associated with overlying scalp infections/inflammation will not be injected. Each catheter will be gently aspirated after the Rickham has been accessed but prior to M032 inoculation; catheters from which CSF can be aspirated will not be inoculated to avoid inoculation into the CSF space. The MRI obtained immediately prior to assessment (see schedule, below) will be used to help inform the decision-making above. If there is any question regarding reservoir/catheter suitability, an additional CT or MRI may be obtained prior to inoculation at the PI's discretion.

Combined Pembrolizumab and M032 treatments at each dose level will be repeated at three-week intervals for up to three cycles total, or until unacceptable toxicity or tumor progression occurs. Patients who are responding to treatment may be considered for additional dosing after the trial period has been completed.

The first two patients treated will not require any waiting period between enrollments. If one of the two should develop a toxicity, the third and subsequent (up to six) patients at that level will not be enrolled until seven weeks from the initial dose of M032 and three weeks from the first combined dose of Pembrolizumab and M032 has transpired for the initial two patients and every patient thereafter, to allow adequate duration of time for development of potential dose limiting toxicities in each treated patient before treating the next patient at that level.

Patients will undergo and then subsequently with each dose of Pembrolizumab; i If one toxicity occurs at a given dose level, that cohort will be increased to 6 patients. If 2 or more toxicities occur at the tested dose level, then with the approval of the DSMB, the dose will be de-escalated by one log and a new cohort enrolled with similar rules at the level. If 2 or more toxicities occur at the deescalated dose level, then the DSMB will be consulted to determine if a stopping rule should be invoked or consideration of further dose de-escalation should be considered. The investigators anticipate as few as four patients (given two or more DLTs initially) and as many as 12 (only one DLT at each dose level). However, based on experience with M032 and Pembrolizumab, the investigators expect that this combination will not produce any dose-limiting toxicities (DLTs).

Phase II: Having established for the safety and tolerability of M032 in conjunction with Pembrolizumab in patients with newly-diagnosed MG, the trial will immediately transition into a Phase II study of Pembrolizumab and M032 in patients with newly diagnosed MG. Patients who are previously untreated but suspected of having a high grade glioma by MRI and are eligible for craniotomy and resection will be offered participation in this two-Cohort trial. Unlike the Phase I, patients will be eligible to receive Pembrolizumab and M032 every 3 weeks for up to one year. The Phase II design will employ the Simon two-stage optimal study design. It will be a single-arm open-label study of M032+ pembrolizumab and the primary endpoints of Over-all Survival at 12 months and 24 months, and Progression Free Survival rate at 6 months (PFS-6). In the first stage, 6 patients will be accrued. Data will be allowed to mature, and an interim analysis per-formed at that time. During this period, additional subjects may be accrued. If there are 2 or fewer responses in the initial 6 patients, further accrual to the study may be stopped. Otherwise, 10 additional patients will be accrued for a total of 16. The null hypothesis will be rejected if 11 or more responses are observed in 16 patients. This design yields a type I error rate of 0.05 and power of 80% when the PFS-6 is 75%. To allow for 25% unevaluable subjects, a maximum of 22 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

Phase I/Cohort I: Participants are eligible to be included in the study only if all of the following criteria apply:

Patients must have histologically or cytologically confirmed glioblastoma multiforme, anaplastic astrocytoma, or gliosarcoma, and is deemed a potential candidate for resection of the recurrent tumor.

Prior therapy: Patients must have failed external beam radio-therapy to the brain, and if eligible and tolerated, undergone appropriate treatment with temozolomide chemotherapy. All radiation and additional chemotherapies must have been completed at least 4 weeks prior to enrollment. Prior therapy with nitrosoureas must have been completed at least 6 weeks prior to enrollment.

Phase I/Cohort II or Phase II: Participants are eligible to be included in the study only if all of the following criteria apply:

Patient must have MRI findings consistent with probable malignant glioma, have no previous diagnosis of glioma, and have had either no history of any surgery for brain tumor. The exception to this requirement is that patients who have under-gone biopsy for diagnosis only and have not received any other treatment. All patients must be potential candidates for resection of the probably malignant glioma tumor.

Should a patient in Phase I/Cohort II or Phase II be found on final pathologic diagnosis to not have a glioblastoma multiforme, anaplastic astrocytoma, or gliosarcoma, he/she will receive no other doses of M032 other than that administered at the time of craniotomy, nor will he/she receive any doses of Pembrolizumab. He/she will be followed for evidence of toxicity of M032 only and will be considered off-study for all efficacy and other secondary endpoints.

All patients, whether in Phase I/Cohort II or Phase II shall also be required to meet the following eligibility and be subject to the exclusion criteria below:

1. Age ≥18 years. Because no dosing or adverse event data are currently available on the use of M032 in patients <16 years of age, children are excluded from this study but will be eligible for future pediatric phase 1 single-agent trials.
2. Karnofsky Performance Status (KPS) ≥70% (see Appendix B).
3. Life expectancy of greater than 4 weeks.
4. Preoperatively, the lesion must be ≥1.0 cm in diameter as determined by MRI.
5. The effects of M032 on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for six months after receiving the final dose of M032. Because it is currently unknown if M032 can be transmitted by sexual contact, a barrier method of birth control must be employed and for six (6) months following the administration of the last dose of this study drug. Should a woman become pregnant while participating in this study, she should inform her treating physician immediately. Subjects should also refrain from donating blood during the trial.
6. Ability to understand and the willingness to sign a written informed con-sent document.
7. Females of childbearing potential must not be pregnant; this will be con-firmed by a negative serum pregnancy test within 14 days prior to starting study treatment.
8. Patients must have normal organ and marrow function as defined below:

   1. leukocytes……………………. >3,000/μl
   2. absolute neutrophil count………. >1,500/μl
   3. platelets…………………………... >100,000/μl
   4. total bilirubin……………………. within normal institutional limits
   5. AST(SGOT)/ALT(SGPT)………… <2.5 X institutional upper limit of normal creatinine within normal institutional limits Or
   6. creatinine clearance……………... >60 mL/min/1.73 m2 for patients with creatinine levels above insti-tutional normal

      Exclusion Criteria:

      A Woman of Child Bearing Potential (WOCBP) who has a positive urine pregnancy test within 72 hours prior to allocation.(see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

      Has received prior therapy with an anti-PD-1, anti-PD-L1, or antiPDL2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX40, CD137).

      Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to allocation.

      Note: Participants must have recovered from all adverse events (AEs) due to previous thera-pies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.

      Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.

      Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.

      Is currently participating in or has participated in a study of an interventionally-directed investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

      Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent or if the agent is directed at analysis and not treatment (e.g., certain PET tracers, etc.).

      Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 2 mg daily of dexamethasone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.

      Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.

      Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.

      Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pitu-tary insufficiency, etc.) is not considered a form of systemic treatment.

      Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.

      Has an active infection requiring systemic therapy.

      Has a known history of Human Immunodeficiency Virus (HIV).

      Has a known history of Hepatitis B (defined as Hepatitis B surface anti-gen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.

      Has a known history of active Bacillus Tuberculosis (TB).

      Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

      Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

      Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening vis-it through 120 days after the last dose of trial treatment.

      Patients who have had chemotherapy, cytotoxic therapy, immunotherapy within 4 weeks prior to entering the study (6 weeks for nitrosoureas), surgical resection within 4 weeks prior to entering the study, or have received experimental viral therapy or gene therapy at any time (e.g., adenovirus, retrovirus or herpes virus protocol). However, this does not preclude re-treatment with M032 at a later date.

      Patients who have not recovered from adverse events due to therapeutic interventions administered more than 4 weeks earlier.

      History of allergic reactions attributed to compounds of similar biologic composition to M032 or to IL-12.

      Tumor involvement which would require ventricular, brainstem, basal ganglia, or posterior fossa inoculation or would require access through a ventricle in order to deliver treatment.

      History of encephalitis within the past 5 years, any history of multiple sclerosis or other CNS infection. Bacterial infections associated with previous cranial operations such as bone flap infections, cerebral abscesses, etc., that have been completely treated will not be exclusions for this trial

      For Phase I, Cohort I: Required steroid increase within 2 weeks of scheduled M032 administration. All study candidates: When possible, the patient should be on a dexamethasone equivalent dose of ≤ 2mg daily at the time of treatment.

      Active herpes lesion.

      Concurrent therapy with any drug active against HSV (acyclovir, valacyclovir, penciclovir, famciclovir, ganciclovir, foscarnet, cidofovir).

      Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or any other medical condition that precludes surgery.

      Patients with known history of allergic reaction to IV contrast material that is not amenable to pre-treatment by protocol.

      Patients with pacemakers, ferro-magnetic aneurysm clips, metal infusion pumps, metal or shrapnel fragments or certain types of stents.

      Receipt of Gliadel Therapy.

      Receipt of Bevacizumab (Avastin) therapy within 4 weeks of scheduled M032 administration. (Receipt of Bevacizumab (Avastin) greater than 4 weeks of scheduled M032 administration does not exclude patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-02-25 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival at 12 and 24 months | 12-24 months
  Overall Survival at 12 and 24 months allows for a quantifiable outcome that should be straightforward to compare to historical data in this patient population.
Progression Free Survival at 6 months (PFS-6) | 6 months
  PFS-6 evaluates all treated patients at 6 months after baseline MRI and determines the percentage of patients who have not progressed by either imaging or neurologic evaluation. The iRA-NO criteria will be utilized to determine progression for this trial. PFS-6 will also be compared to historical controls for each cohort.
Overall Survival (OS) | 3 years
  OS will be determined for each cohort of patients and compared to historical controls for that cohort. .
Progression Free Survival (PFS) | 3 years
  PFS will be determined by MRI and neurologic evaluation using the iRANO criteria. PFS utilizes an historical approach to determining if progression has occurred and is helpful measure to compare this current study to historical studies. An important limitation in the assessment of PFS centers on the fact that patients may not get imaging or neurologic examinations done at an optimal or consistent time; as such, another approach, PFS-6, has been adopted in some studies. PFS-6 evaluates all treated patients at 6 months after baseline MRI and determines the percentage of patients who have not progressed by either imaging or neurologic evaluation. The iRANO criteria will be utilized to determine progression for this trial. PFS and OS will be compared to historical controls for each cohort.

CONTACTS AND LOCATIONS:
Overall Officials: James Markert, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No